CLINICAL TRIAL: NCT06083974
Title: Retrospective Study of Metastatic Left Colon and Rectal Cancer as Regard Treatment With Anti_EGFR Targeted Therapy
Brief Title: Metastatic Left Colon and Rectal Cancer Treatment With Anti_EGFR Targeted Therapy
Acronym: EGFR
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ebrahim mohammed, Principal investigator1, Assiut University
Other Study IDs: Anti_EGFR -Targeted therapy
Record Dates: First submitted 2023-10-04; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Colorectal Adenocarcinoma
Keywords: EGFR, Targeted therapy ,metastatic colorectal cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer ranks the second lethal cancer and third prevalent malignant tumour worldwide, Despite of different odern modalities for diagnosis,large number of cases diagnosed at metastatic advanced stage .

New treatment approach has been discovered habe been discovered making a huge revolution in metastatic colorectal cancer represented by targeted therapy including anti_EGFR ,anti_angiogenic and kinase inhibitors .

DETAILED DESCRIPTION:
Retrospective study aims to evaluate the effect of EGFR expression in metastatic colorectal cancer and the outcome of treatment with anti_EGFR targeted therapy between left colon and rectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. age above 18
2. Both sex
3. Performance status zero to one according to ECOG scale system
4. Histo-pathologial diagnosis adenocarcinoma of left colon or rectum.
5. Patients diagnosed with left colon and rectal cancer.
6. Patients eligible to receive chemotherapy (with renal and liver chemistry, and normal CBC.
7. Patients diagnosed with metastatic stage.
8. K-RAS wild type.

Exclusion Criteria:

1. Second malignancy
2. Histo-pathological types other than adenocarcinoma.
3. Right colon cancer patients.
4. Patients refused receiving anti_EGFR targeted therapy.
5. Patients with any abnormalities preventing to receive chemotherapy.
6. Early stages of colorectal cancer.
7. K-RAS mutant type.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left colon and rectum cancer of stage four received target therapy anti_EGFR targeted therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
OS and DFS of patients with metastatic colorectal cancer patients received anti_EGFR targeted therapy | Anti_EGFR targeted therapy in assuit university hospitals from 2015 to 2022
  Evaluation of anti-EGFR targeted therapy on metastatic cancer rectum and left colon and factors affecting response to treatment

SECONDARY OUTCOMES:
Response rate (RR) in patients received chemotherapy only or with combination with targeted therapy. | The response of patients to EGFR targeted therapy in AUH at period from 2015 to 2022
  Factors affecting response to targeted therapy

CONTACTS AND LOCATIONS:
Overall Officials: Samir E Shehata, Professor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Efficacy and safety of bevacizumab plus chemotherapy in Chinese patients with metastatic colorectal cancer: a randomized phase III ARTIST trial — https://pubmed.ncbi.nlm.nih.gov/21959045/
- See also: Panitumumab-FOLFOX4 treatment and RAS mutations in colorectal cance — https://pubmed.ncbi.nlm.nih.gov/24024839/
- See also: tion between tumour response to first-line chemotherapy and survival in advanced colorectal cancer: a meta-analysis. Meta-Analysis Group in Cancer — https://pubmed.ncbi.nlm.nih.gov/10972369/
- See also: The biology of VEGF and its receptor — https://pubmed.ncbi.nlm.nih.gov/12778165/
- See also: Advances and new perspectives in the treatment of metastatic colon cancer — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4092338/